CLINICAL TRIAL: NCT01620827
Title: Study Subject Responsiveness to Follow-Up Phone Calls From a Hospital Landline as Compared With From a Private Cellular Phone Number
Brief Title: Hospital vs. Cell Phone Number Follow-Up Randomization Study
Acronym: FURS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HUP-FURS-2012
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Subject Follow-up
Keywords: follow up; cell phone; hospital landline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hospital Landline (Active Comparator): Subjects in this arm have all of their follow-up phone calls placed from a hospital landline number.
  Interventions: Other: Hospital Landline Phone Calls
- Private Cell Phone (Active Comparator): Subjects in this arm have all of their follow-up phone calls placed from a private cell phone number.
  Interventions: Other: Private Cell Phone Calls

INTERVENTIONS:
Other: Hospital Landline Phone Calls — Follow-up phone calls are made from the hospital landline phones in a research office
  Arms: Hospital Landline
Other: Private Cell Phone Calls — Follow-up phone calls are made from the private cell phones of research assistants
  Arms: Private Cell Phone

SUMMARY:
This study is being conducted to evaluate the hypothesis that study subjects will be more responsive to follow-up phone calls made from personal cell phone numbers than from hospital landline numbers. To evaluate this, study subjects previously enrolled in a cardiac biomarker study (the Early Identification of Acute Coronary Syndrome study) were randomized to receive their follow-up phone calls (the calls associated with the Early ID study occur at 30 days and 1 year after initial enrollment) from either a hospital office landline or from the personal cell phones of the research assistants making these calls. This was done as a 1:1 randomization. The number of call attempts required to reach the study subjects were recorded as the calls were made and the date of successful follow-up was recorded once contact was made.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the Early Identification of Acute Coronary Syndrome study
* Working telephone numbers

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Successful phone call contact at 30 days | 90 days
  Contact is attempted from 30 days after enrollment through 90 days after enrollment. If contact is made during this time frame, 30 day follow-up is considered to have been successful.

SECONDARY OUTCOMES:
The number of call attempts required to obtain successful follow-up | 90 days
  Contact is attempted from 30 days after enrollment through 90 days after enrollment. The number of calls required to make successful contact in this time frame are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Judd Hollander, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States